CLINICAL TRIAL: NCT06009250
Title: Prevalence of Non-alcoholic Fatty Liver Disease in Patients With Chronic Kidney Disease in Assiut
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Muhammad Ameen Abdelrady Abdelaziz (Other)
Responsible Party: Sponsor-Investigator, Muhammad Ameen Abdelrady Abdelaziz, Internal Medicine Resident, Assiut University
Organization: Assiut University (Other)
Other Study IDs: NAFLD and CKD
Record Dates: First submitted 2023-07-28; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: CKD; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- CKD patients: CKD patient who are not DM are investigated for the presence of NAFLD
- normal control group: normal population are investigated to know the prevalence of NAFLD in contrast to patients with CKD.

SUMMARY:
The goal of this observational study is to detect the prevalence of NAFLD in CKD patients

The main question[s] it aims to answer are:

* [question 1] prevalence of NAFLD in CKD patients.
* [question 2] the relationship between NAFLD and CKD.

DETAILED DESCRIPTION:
The goal of this observational study is to detect the prevalence of NAFLD in CKD patients

The main question[s] it aims to answer are:

* [question 1] prevalence of NAFLD in CKD patients.
* [question 2] the relationship between NAFLD and CKD.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients

Exclusion Criteria:

* HCV and HBV Positive patients
* Alcoholics
* patient on Hemodialysis
* patients with wilson disease
* patients with alpha one antitrypsin deficiency

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: CKD patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
abdominal ultrasound | 1 year
  assessment of Liver regarding fatty liver disease by Ultrasound.
liver enzymes | 1 year
  participants will undergo assessment of liver enzymes (AST and ALT) and results will be reporeted in a table.
Fibroscan | 1 year
  participants will undergo fibroscanning of the liver to assess NAFLD and results will be reported in a table.
BUN, Cr level and estimated GFR | 1 year
  participants will be assessed regarding BUN, CR and estimated GFR to confirm and follow up CKD patients involved in the study.
Lipid Profile | 1 year
  participants will be assessed regarding Cholesterol level, Triglycerides, HDL and LDL. results will be reported in a table
Complete Blood Picture (WBCs, HB, Patelets | 1 year
  total leucocytic count Hemoglobin level and platelet count will be assessed in our patients and will be reported in a table
serum Uric Acid | 1 year
  serum uric acid will be assessed and reported in our patients

SECONDARY OUTCOMES:
Waist Circumference | 1 year
  waist circumference measurement.
Body Mass Index | 1 year
  BMI will also be calculated.